CLINICAL TRIAL: NCT01810900
Title: To Assess the Anti-adhesive Effect and Safety of Protescal Following Laparoscopic Surgery
Brief Title: To Assess the Anti-adhesive Effect and Safety of Protescal
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LG-ABCL002
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2014-11

CONDITIONS: Laparoscopic Myomectomy
Keywords: anti-adhesive effect and safety, laparoscopic myomectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protescal (Experimental): Protescal is applied to this arm.
  Interventions: Device: Protescal
- non-treatment (No Intervention)

INTERVENTIONS:
Device: Protescal
  Arms: Protescal

SUMMARY:
This multicenter, randomized, single-blind study assessed the safety and efficacy of Protescal for the reduction of post-operative adhesion formation following myomectomy.

DETAILED DESCRIPTION:
The age of the patients participating in the study overed 20 years and included nonpregnant women requiring laparoscopic myomectomy and expected to undergo a second-look laparoscopy as part of their treatment plan 5 weeks after the initial surgery.

ELIGIBILITY:
Inclusion Criteria:

* a woman who is over 20 years old
* a woman who needs a laparoscopic myomectomy

Exclusion Criteria:

* a pregnant woman and a nursing mother

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
presence/absence of postoperative adhesions at second-look procedure | at second look laparoscopy after 5 weeks later initial laparoscopic myomectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Hospital, Seoul, Seoul, South Korea